CLINICAL TRIAL: NCT03180827
Title: Female Fertility Preservation Using Ovarian Tissue Cryopreservation Before Highly Gonadotoxic Cancer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gumy-Pause Fabienne (Other)
Responsible Party: Sponsor-Investigator, Gumy-Pause Fabienne, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PB_2017-00536 (15-073)
Record Dates: First submitted 2017-05-31; First posted 2017-06-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Childhood Cancer; Fertility Disorders
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ovarian tissue cryopreservation (Experimental)
  Interventions: Procedure: ovarian tissue biopsy

INTERVENTIONS:
Procedure: ovarian tissue biopsy — ovarian tissue biopsy during general anesthesia

SUMMARY:
Background:

Due to the remarkable improvement in treatments these last decades, long term survival can be expected in more than 80% of childhood cancer patients. Unfortunately, cancer treatments can be harmful to the gonads and can affect reproductive and endocrine functions. While loss of fertility is a major concern for most patients, only the experimental option of ovarian tissue cryopreservation can be proposed to prepubertal girls with a high risk of infertility. For pubertal patient, cryopreservation of mature oocytes after ovarian stimulation can be offered if oncological treatment debut can be delayed. As it is often not possible, ovarian tissue cryopreservation can also be offered.

Primary aims

- To cryopreserve ovarian tissue of pre or peripubertal patient who will be receiving highly gonadotoxic oncological treatment.

Secondary aims

* To create a database in order to record clinical and biological follow-up data
* To pool resources with Fertisave Registry
* To create a research biobank for future research projects

Multicentric study: HUG, CHUV

ELIGIBILITY:
Inclusion Criteria:

* Pediatric pre ou peripubertal patient aged 2 months and older
* Patient presenting high risk of infertility because of gonadotoxic treatments (i.e. high dose of alkylating agents, ovarian irradiation, total body irradiation)
* Multidisciplinary team consensus in favour to proposition to cryopreserve ovarian tissue.

Exclusion Criteria:

* Patient under the age of 2 months
* Refusal of the patient and/or her parents
* Treatments that are not highly gonadotoxic

Ages: 2 Months to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2100-01 (Estimated); Study Completion 2100-01 (Estimated)

PRIMARY OUTCOMES:
Number of pediatric cancer patient who will undergo ovarian tissue cryopreservation for fertility preservation | 0-20 years

SECONDARY OUTCOMES:
Incidence of complications related to the ovarian biopsy (safety) | 0-20 years
  The safety will be assessed by recording the number of complications of the procedure (e.g. bleeding, infection)
Comparison of biochemical markers | 0-20 years
  Comparison of biochemical markers (e.g., FSH; LH, AMH, progesterone, oestradiol) between patients who undergo ovarian biopsy and controls

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Gumy-Pause, Dr, Study Chair — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - Geneva University Hospitals, Geneva
  - CHUV, Lausanne